CLINICAL TRIAL: NCT04088799
Title: Effect of LDL-Apheresis on Cardiovascular and Renal Outcomes in Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: LDL-Apheresis for FSGS CardioRenal Outcomes
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CIN001 - LDL Outcomes
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples from before and after LDL apheresis treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FSGS requiring LDL-apheresis: Pediatric patients with FSGS requiring LDL-apheresis with the Liposorber
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Focal segmental glomerulosclerosis (FSGS) is the most common cause of end-stage renal disease (ESRD) in adolescents. The refractory nature of FSGS and a more than 30% recurrence rate after kidney transplantation renders treatment of FSGS one of the most difficult challenges in pediatric nephrology. A significant knowledge gap in understanding the mechanism of FSGS treatment resistance and progression hampers development of successful treatment strategies. Beneficial effect of removal of low-density lipoproteins by LDL-apheresis indicates that lipids contribute to progression in FSGS.

The investigators will test the hypothesis that removal of Lp-PLA2 and lipid metabolites by LDL-apheresis ameliorates proteinuria and cardiovascular comorbidities. Patients with FSGS and FSGS recurrence after kidney transplantation receiving LDL-apheresis as part of standard of care will be enrolled to the study. Pre-and post serum and effluent concentrations of LPC, free FA, Lp-PLA2, oxidized LDL, fasting lipid profile, interleukin (IL)-6, tumor necrosis factor (TNF)-α, and IL-1β will be monitored in patients undergoing LDL-apheresis. Investigators will also study the impact of LDL-apheresis on cardiovascular and clinical comorbidities by monitoring degree of proteinuria, blood pressures and arterial stiffness index.

DETAILED DESCRIPTION:
Focal segmental glomerulosclerosis (FSGS) is the most common cause of end-stage renal disease (ESRD) in adolescents. The refractory nature of FSGS and a more than 30% recurrence rate after kidney transplantation renders treatment of FSGS one of the most difficult challenges in pediatric nephrology. A significant knowledge gap in understanding the mechanism of FSGS treatment resistance and progression hampers development of successful treatment strategies. Beneficial effect of removal of low-density lipoproteins by LDL-apheresis indicates that lipids contribute to progression in FSGS. We have previously reported increased urinary fatty acids (FA) and lysophosphatidylcholines (LPC) levels with non-targeted urinary lipidomic analysis in children with FSGS. Unregulated phospholipase A2(PLA2) activity causes an increase in intracellular concentrations of free FA and LPC altering plasma membrane and mitochondrial permeability.

Lipoprotein associated PLA2 is a biomarker involved in oxidative modification of LDL by hydrolyzing oxidative lysophosphatidylcholines (LPC) and oxidized free fatty acids (FFA) both of which are proinflammatory and atherogenic. Lp-PLA2 is efficiently removed by LDL-apheresis. The investigators hypothesize that LDL-apheresis ameliorates cellular injury and vascular changes by removing circulating Lp-PLA2, oxidized LDL, LPC, FA and cytokines in FSGS. In this proposal, the hypothesis that removal of Lp-PLA2 and lipid metabolites by LDL-apheresis ameliorates proteinuria and cardiovascular comorbidities will be tested. Patients with FSGS and FSGS recurrence after kidney transplantation receiving LDL-apheresis as part of standard of care will be enrolled to the study. Investigators will monitor pre-and post serum and effluent concentrations of LPC, free FA, Lp-PLA2, oxidized LDL, fasting lipid profile, IL-6, TNF-α, and IL-1β of patients undergoing LDL-apheresis. The impact of LDL-apheresis on cardiovascular and clinical comorbidities by monitoring degree of proteinuria, blood pressures and arterial stiffness index will also be investigated.

The investigators propose that LDL-apheresis as a conjunct therapy to standard treatment regimens is an efficient way to ameliorate progression prevent comorbidities such as systemic inflammation and lipid induced vascular changes thus progression in FSGS. Furthermore, removal of Lp-PLA2 and other lipids by LDL-apheresis can limit the direct toxicity caused by lipid metabolites to podocytes and proximal tubule epithelial cells. The investigators believe that this proposal will enhance understanding of lipid-mediated progression in FSGS and will delineate the role of LDL-apheresis as part of established treatment in treatment of FSGS.

ELIGIBILITY:
Inclusion Criteria:

* FSGS and a glomerular filtration rate (GFR) ≥ 60 ml/min/1.73m2 AND

  * Refractory nephrotic syndrome in which standard treatment options are unsuccessful (i.e., patient is unresponsive to standard corticosteroid and/or calcineurin inhibitor therapy for at least 8 weeks resulting in failure to achieve complete or partial remission), OR
  * Refractory nephrotic syndrome in which standard treatment options are not well tolerated (i.e., patients intolerant to standard therapies due to severe side effects without providing an acceptable level of clinical benefit), OR
  * Refractory or recurrent nephrotic syndrome in which standard therapy is contraindicated
* Post renal transplant with nephrotic syndrome associated with primary FSGS

Exclusion Criteria:

* Greater than 21 years of age
* Parent or patient unwilling or unable to signed and date the informed consent
* Pregnant, lactating, or planning to become pregnant prior to completing the study
* Unable or unwilling to comply with the follow-up schedule
* Simultaneously participating in another investigational drug or device study (except for LDL-apheresis associated trials)
* Body weight less than 21 kilograms (46 pounds)
* Currently being administered angiotensin converting enzyme (ACE) inhibitors that cannot be withheld for at least 24 hours prior to each apheresis treatment
* Currently being administered antihypertensive drugs other than ACE inhibitors than cannot be withheld on the day of LDL-apheresis until after the procedure
* Medical condition or disorder that would limit life expectancy to less than the primary clinical study endpoint or that may cause noncompliance with the study plan or confound the data analysis
* Hypersensitivity to dextran sulfate, heparin, or ethylene oxide
* Inability to achieve adequate anticoagulation
* Inability to tolerate extracorporeal circulation therapy with Liposorber® LA-15
* Cardiac impairments such as uncontrolled arrhythmia, unstable angina, decompensated congestive heart failure, or valvular disease
* Thyroid disease or liver abnormalities
* Unresolved systemic or local infection that could affect the clinical study outcomes

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with focal segmental glomerulosclerosis (FSGS) in need of LDL-apheresis per standard of care
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Severity of Proteinuria | 9 weeks
  Standard of care proteinuria will be monitored for expected improvement in severity

SECONDARY OUTCOMES:
Cardiovascular comorbidities | 9 weeks
  LPC, free FA, Lp-PLA2, oxidized LDL, IL-6, TNF-α, and IL-1β will be monitored from patient blood before and after and from the effluent at LDL-apheresis treatments

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No